CLINICAL TRIAL: NCT01622569
Title: A 16-Week Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study Evaluating the Efficacy and Safety of Intranasal Administration of 100, 200, and 400 μg of Fluticasone Propionate Twice a Day (BID) Using a Novel Bi Directional Device in Subjects With Bilateral Nasal Polyposis Followed by an 8-Week Open-Label Extension Phase to Assess Safety
Brief Title: Study Evaluating the Efficacy and Safety of Intranasal Administration of 100, 200, and 400 μg of Fluticasone Propionate Twice a Day (BID) Using a Novel Bi Directional Device in Subjects With Bilateral Nasal Polyposis Followed by an 8-Week Open-Label Extension Phase to Assess Safety
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Optinose US Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPN-FLU-NP-3101
Record Dates: First submitted 2012-06-13; First posted 2012-06-19 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2017-11

CONDITIONS: Bilateral Nasal Polyposis
MeSH Terms: interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- OPN-375 100 μg BID (Active Comparator): Double-Blind Treatment Phase: OPN-375 100 μg BID x 16 weeks
  Open-Label Extension Phase: OPN-375 400 μg BID x 8 weeks
  Interventions: Drug: Fluticasone Propionate
- Placebo (Placebo Comparator): Double-Blind Treatment Phase: Matching Placebo BID x 16 weeks
  Open-Label Extension Phase: OPN-375 400 μg BID x 8 weeks
  Interventions: Drug: Fluticasone Propionate
- OPN-375 200 μg BID (Active Comparator): Double-Blind Treatment Phase: OPN-375 200 μg BID x 16 weeks
  Open-Label Extension Phase: OPN-375 400 μg BID x 8 weeks
  Interventions: Drug: Fluticasone Propionate
- OPN-375 400 μg BID (Active Comparator): Double-Blind Treatment Phase: OPN-375 400 μg BID x 16 weeks
  Open-Label Extension Phase: OPN-375 400 μg BID x 8 weeks
  Interventions: Drug: Fluticasone Propionate

INTERVENTIONS:
Drug: Fluticasone Propionate — Delivered via Optinose Exhalation Delivery System
  Other Names: OPN-375

SUMMARY:
The primary objective of this study is to compare the efficacy of intranasal administration of 100, 200, and 400 μg of fluticasone propionate twice a day delivered by the OptiNose device with placebo in subjects with bilateral nasal polyposis. Two co-primary endpoints will be used in the study: reduction of nasal congestion/obstruction symptoms at the end of Week 4 of the double-blind treatment phase measured by the 7 day average instantaneous AM diary symptom scores, and reduction in total polyp grade (sum of scores from both nasal cavities) over the 16 weeks of the double-blind treatment phase as determined by the Lildholdt scale score measured by nasoendoscopy.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled, parallel-group, multicenter study designed to assess the efficacy and safety of intranasal administration of 3 doses of OPN-375 (100, 200, and 400 µg bid) in subjects with bilateral nasal polyposis and nasal congestion.

This study consisted of 3 phases. After signing informed consent, subjects who met eligibility criteria at Visit 1 (screening) entered the study.

1. Pretreatment phase (single-blind, placebo, run-in): 7 to up to 14 days duration, to determine disease status eligibility and to ensure the subject was able to comply with study procedures prior to randomization and enrolment in the double-blind treatment phase.
2. Double-blind treatment phase: 16 weeks duration with 6 scheduled visits starting with Visit 2, Day 1 (baseline) when eligible subjects were randomized by balance allocation to 1 of 4 treatment groups and ending at Visit 7 (Week 16).
3. Open-label extension phase: 8 weeks duration with 1 scheduled visit (Visit 8 [Week 24]).

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 years and older
* Women must

  * be practicing an effective method of birth control (eg,prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double-barrier method [eg, condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel], or male partner sterilization) before entry and throughout the study, or
  * be surgically sterile (have had a hysterectomy or bilateral oophorectomy, or tubal ligation at least 1 year before screening) or otherwise be incapable of pregnancy, or
  * be postmenopausal (spontaneous amenorrhea for at least 1 year).
* Women of child-bearing potential must have a negative serum beta-human chorionic gonadotropin (B-hCG) or urine pregnancy test (depending on local regulations) at the screening visit
* Must have bilateral nasal polyposis with a grade of 1 to 3 in each of the nasal cavities as determined by the Lildholdt scale score measured by nasoendoscopy at both screening and baseline visits
* Must have at least moderate symptoms of nasal congestion/obstruction as reported by the subject for the 7 day period preceding the screening visit
* At the baseline visit (Day 1), must have a morning score of at least 2 (moderate) on nasal congestion/obstruction recorded on the subject diary for at least 5 of the last 7 days of the 7 to up to 14 day run-in period
* Must demonstrate an ability to correctly complete the daily diary during the run-in period to be eligible for randomization
* Subjects with comorbid asthma or COPD must be stable with no exacerbations (eg, no emergency room visits, hospitalizations, or oral or parenteral steroid use) within the 3 months before the screening visit. Inhaled corticosteroid use must be limited to stable doses of no more than 1,000 μg/day of beclomethasone (or equivalent) for at least 3 months before screening with plans to continue use throughout the study.
* Must be able to cease treatment with intranasal medications including, but not limited to, intranasal steroids, intranasal sodium cromolyn, nasal atropine, nasal ipratropium bromide, inhaled corticosteroids (except permitted doses listed above for comorbid asthma and COPD) at the screening visit
* Must be able to cease treatment with oral and nasal decongestants and antihistamines at the screening visit
* Must be able to use the OptiNose device correctly; all subjects will be required to demonstrate correct use of the placebo device at screening, Visit 1.
* Must be capable, in the opinion of the investigator, of providing informed consent to participate in the study. Subjects must sign an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* Women who are pregnant or lactating
* Have complete or near-complete obstruction of the nasal cavities
* Inability to achieve bilateral nasal airflow for any reason including nasal septum deviation
* Inability to have each nasal cavity examined for any reason including nasal septum deviation
* Nasal septum perforation
* Has had more than 1 episode of epistaxis with frank bleeding in the month before the screening visit
* Have evidence of significant baseline mucosal injury, ulceration or erosion (eg, exposed cartilage, perforation) on baseline nasal examination/nasal endoscopy
* History of more than 5 sinonasal surgeries for either nasal polyps or nasal/sinus inflammation (lifetime)
* History of sinus or nasal surgery within 6 months before the screening visit
* History of any surgical procedure that prevents the ability to accurately grade polyps
* Have symptoms of seasonal allergic rhinitis at screening or baseline and/or, based on time of year, would anticipate onset of symptoms within 4 weeks of randomization
* Current, ongoing rhinitis medicamentosa (rebound rhinitis)
* Have significant oral structural abnormalities, eg, a cleft palate
* Diagnosis of cystic fibrosis
* History of Churg-Strauss syndrome or dyskinetic ciliary syndromes
* Purulent nasal infection, acute sinusitis, or upper respiratory tract infection within 2 weeks before the screening visit. Potential subjects presenting with any of these infections may be rescreened 4 weeks after symptom resolution Note: Subjects who are taking prophylactic antibiotics will be allowed to enter the study as long as they intend to continue the antibiotics for the duration of the study.
* Planned sinonasal surgery during the period of the study
* Allergy, hypersensitivity, or contraindication to corticosteroids or steroids
* Allergy or hypersensitivity to any excipients in study drug
* Exposure to any glucocorticoid treatment with potential for systemic effects (eg, oral, parenteral, intra-articular, or epidural steroids, high dose topical steroids) within 1 month before the screening visit; except as noted in inclusion criteria for subjects with comorbid asthma or COPD
* Have nasal candidiasis
* Have taken a potent CYP3A4 inhibitor within 14 days before the screening visit.
* History or current diagnosis of any form of glaucoma or ocular hypertension (ie, >21 mmHg)
* History of intraocular pressure elevation on any form of steroid therapy
* History or current diagnosis of the presence (in either eye) of a cataract
* Any serious or unstable concurrent disease, psychiatric disorder, or any significant condition that, in the opinion of the investigator could confound the results of the study or could interfere with the subject's participation or compliance in the study
* A recent (within 1 year of the screening visit) clinically significant history of drug or alcohol use, abuse, or dependence that, in the opinion of the investigator could interfere with the subject's participation or compliance in the study
* Positive urine drug screen at screening visit for drugs of abuse, with the exception of prescribed medications for legitimate medical conditions
* Have participated in an investigational drug clinical trial within 30 days of the screening visit
* Employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2013-11-19 (Actual); Primary Completion 2015-08-06 (Actual); Study Completion 2015-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (30):
  - SC Clinical Research, Inc., Tucson, Arizona
  - Kern Allergy and Medical Research, Inc., Bakersfield, California
  - Central California Clinical Research, Fresno, California
  - Allergy & Asthma Specialists Medical Group, Huntington Beach, California
  - California Allergy & Asthma Medical Group, Inc., Los Angeles, California
  - Choc PSF, AMC, Division of AA & I, Orange, California
  - California Allergy and Asthma Palmdale, Palmdale, California
  - Peninsula Research Associates, Inc., Rolling Hills Estates, California
  - California Medical Clinic for Headache, Santa Monica, California
  - Asthma & Allergy Associates, P.C., Colorado Springs, Colorado
  - Colorado ENT & Allergy, Colorado Springs, Colorado
  - Colorado Allergy and Asthma Centers, P.C., Denver, Colorado
  - University of South Florida Asthma, Allergy & Immunology, Tampa, Florida
  - NU Feinberg School of Medicine Depart. of Otolaryngology-Head & Neck Surgery, Chicago, Illinois
  - Chicago ENT, Chicago, Illinois
  - Northeast Medical Research Associates, Inc, North Dartmouth, Massachusetts
  - The Center for Pharmaceutical Research, P.C., Kansas City, Missouri
  - Clinical Research Group of Montana, PLLC, Bozeman, Montana
  - Coastal Ear, Nose and Throat, LLC, Neptune City, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Optimed Research, Columbus, Ohio
  - Allergy, Asthma & Clinical Research Center, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, Tulsa, Oklahoma
  - National Allergy, Asthma & Urticaria Centers of Charleston, P.A., North Charleston, South Carolina
  - AARA Research Center, Dallas, Texas
  - Ear Nose and Throat Associates of Texas, Frisco, Texas
  - ENTTEX, Plano, Texas
  - EVMS Depart. Of Otolaryngology, Norfolk, Virginia
  - Allergy, Asthma & Sinus Center, S.C., Greenfield, Wisconsin
- Canada (3):
  - Ottawa Allergy Research Corporation, Ottawa, Ontario
  - CHUM Hôtel-Dieu, Montreal, Quebec
  - Dr. Jaime Del Carpio, Montreal, Quebec

REFERENCES:
- [Derived] Ow RA, McGinnis JP 2nd, Sacks HJ, Mehle ME. The Effect of EDS-FLU on Objective and Patient-Reported Subjective Outcomes for Patients with Chronic Rhinosinusitis with Nasal Polyps. Ear Nose Throat J. 2025 Feb;104(2):93-101. doi: 10.1177/01455613221088698. Epub 2022 Apr 18. PMID 35437059
- [Derived] Skoner DP, Meltzer EO, Skoner J, Sacks HJ, Lumry WR. Evaluation of the ocular safety associated with the exhalation delivery system with fluticasone. Allergy Asthma Proc. 2022 Jan 9;43(1):70-77. doi: 10.2500/aap.2022.43.210096. Epub 2021 Nov 9. PMID 34753535

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching placebo BID x 16 weeks, then OPN-375 (open-label) 400 μg BID x 8 weeks
- 100 μg OPN-375: OPN-375 100 μg BID x 16 weeks, then OPN-375 (open-label) 400 μg BID x 8 weeks
- 200 μg OPN-375: OPN-375 200 μg BID x 16 weeks, then OPN-375 (open-label) 400 μg BID x 8 weeks
- 400 μg EDS-FLU: OPN-375 400 μg BID x 16 weeks, then OPN-375 (open-label) 400 μg BID x 8 weeks
Period: Double-Blind Treatment Phase (Wks 1-16)
Arm/Group | Placebo | 100 μg OPN-375 | 200 μg OPN-375 | 400 μg EDS-FLU
Started | 82 | 81 | 80 | 80
Completed | 70 | 75 | 71 | 76
Not Completed | 12 | 6 | 9 | 4
Not completed — Adverse Event | 4 | 2 | 3 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 6 | 0 | 3 | 2
Not completed — Protocol Violation | 0 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 2 | 0
Period: Open-Label Extension Phase (Wks 17-24)
Arm/Group | Placebo | 100 μg OPN-375 | 200 μg OPN-375 | 400 μg EDS-FLU
Started | 68 | 72 | 67 | 75
Completed | 67 | 70 | 64 | 73
Not Completed | 1 | 2 | 3 | 2
Not completed — Adverse Event | 0 | 2 | 1 | 0
Not completed — Lack of Efficacy | 1 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Matching Placebo BID x 16 weeks, then OPN-375 400 μg (open-label) BID x 8 weeks
- OPN-375 100 μg BID: OPN-375 100 μg BID x 16 weeks, then OPN-375 400 μg (open-label) BID x 8 weeks
- OPN-375 200 μg BID: OPN-375 200 μg BID x 16 weeks, then OPN-375 400 μg (open-label) BID x 8 weeks
- OPN-375 400 μg BID: OPN-375 400 μg BID x 16 weeks, then OPN-375 400 μg (open-label) BID x 8 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo | OPN-375 100 μg BID | OPN-375 200 μg BID | OPN-375 400 μg BID | Total
Number analyzed (Participants) | 82 | 81 | 80 | 80 | 323
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (13.0) | 44.9 (12.7) | 46.4 (12.7) | 43.9 (12.6) | 45.1 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 41 | 32 | 42 | 161
  Male | 36 | 40 | 48 | 38 | 162
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 68 | 74 | 72 | 69 | 283
  Black/African American | 8 | 3 | 6 | 9 | 26
  Asian | 5 | 2 | 2 | 0 | 9
  Other | 1 | 2 | 0 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 4 | 5 | 5 | 4 | 18
  Czechia | 14 | 15 | 14 | 13 | 56
  United Kingdom | 3 | 2 | 2 | 4 | 11
  Ukraine | 16 | 17 | 16 | 16 | 65
  United States | 36 | 36 | 35 | 36 | 143
  South Africa | 9 | 6 | 8 | 7 | 30
Total Polyp Grading Score (sum of scores from both nasal cavities) [Mean (Full Range); unit: Units on a Scale] — Polyp grading of each nasal cavity was determined by a nasal polyp grading scale score measured by nasoendoscopy.
  0: No polyps
  1. Mild polyposis: polyps not reaching below the inferior border of the middle turbinate
  2. Moderate polyposis: polyps reaching below the inferior border of the middle concha, but not the inferior border of the inferior turbinate
  3. Severe polyposis large polyps reaching below the lower inferior border of the inferior turbinate Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  Included patients with nasal polyps at baseline
  Units on a Scale
    number analyzed (Participants) | 82 | 81 | 80 | 79 | 322
    (all) | 3.8 [2 to 6] | 3.6 [2 to 6] | 3.9 [2 to 6] | 3.7 [2 to 6] | 3.75 [2 to 6]
Use of intranasal corticosteroid (ICS) treatment for polyps in past 10 years [Count of Participants; unit: Participants] | 77 | 77 | 76 | 75 | 305
Previous sinus surgery for polyp removal or sinus surgery [Count of Participants; unit: Participants] — Patients may have had both sinus surgery and polypectomy.
  Participants | 33 | 34 | 27 | 30 | 124
Previous polyp removal surgery via polypectomy only [Count of Participants; unit: Participants] — Patients may have had both sinus surgery and polypectomy.
  Participants | 33 | 27 | 33 | 27 | 120
Nasal Congestion/Obstruction Score (7-Day Instantaneous Morning) [Mean (Full Range); unit: units on a scale] — Subjects reported nasal symptoms using the electronic diary twice daily immediately before dosing.
  0: None
  1. Mild - symptoms clearly present, but minimal awareness, and easily tolerated
  2. Moderate - definite awareness of symptoms that is bothersome but tolerable
  3. Severe - symptoms that are hard to tolerate, cause interference with activities or daily living Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  units on a scale
    number analyzed (Participants) | 82 | 81 | 80 | 79 | 322
    (all) | 2.31 [1.7 to 3.0] | 2.22 [0.8 to 3.0] | 2.24 [1.6 to 3.0] | 2.29 [1.7 to 3.0] | 2.27 [0.8 to 3.0]
Rhinorrhea Score (7-day instantaneous morning) [Mean (Full Range); unit: units on a scale] — Subjects reported nasal symptoms using the electronic diary twice daily immediately before dosing.
  0: None
  1. Mild - symptoms clearly present, but minimal awareness, and easily tolerated
  2. Moderate - definite awareness of symptoms that is bothersome but tolerable
  3. Severe - symptoms that are hard to tolerate, cause interference with activities or daily living Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  units on a scale
    number analyzed (Participants) | 82 | 81 | 80 | 79 | 322
    (all) | 1.81 [0.0 to 3.0] | 1.67 [0.0 to 3.0] | 1.75 [0.0 to 3.0] | 1.83 [0.0 to 3.0] | 1.76 [0.0 to 3.0]
Facial Pain or Pressure Score (7-day instantaneous morning) [Mean (Full Range); unit: units on a scale] — Subjects reported nasal symptoms using the electronic diary twice daily immediately before dosing.
  0: None
  1. Mild - Symptoms clearly present, but minimal awareness, and easily tolerated
  2. Moderate - Definite awareness of symptoms that is bothersome but tolerable
  3. Severe - Symptoms that are hard to tolerate, cause interference with activities or daily living Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  units on a scale
    number analyzed (Participants) | 82 | 81 | 80 | 79 | 322
    (all) | 1.65 [0.0 to 3.0] | 1.53 [0.0 to 3.0] | 1.48 [0.0 to 3.0] | 1.62 [0.0 to 3.0] | 1.57 [0.0 to 3.0]
Hyposomia Score (7-day instantaneous morning) [Mean (Full Range); unit: units on a scale] — Subjects reported nasal symptoms using the electronic diary twice daily immediately before dosing.
  0: None
  1. Mild - Symptoms clearly present, but minimal awareness, and easily tolerated
  2. Moderate - Definite awareness of symptoms that is bothersome but tolerable
  3. Severe - Symptoms that are hard to tolerate, cause interference with activities or daily living Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, an who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  units on a scale
    number analyzed (Participants) | 82 | 81 | 80 | 79 | 322
    (all) | 2.42 [0.0 to 3.0] | 2.31 [0.0 to 3.0] | 2.49 [0.0 to 3.0] | 2.44 [0.0 to 3.0] | 2.41 [0.0 to 3.0]
Sinonasal Outcome Test 22 (SNOT-22) Total Score [Mean (Full Range); unit: units on a scale] — SNOT-22 is a subject-completed questionnaire that consists of 22 questions. The questions on the SNOT-22 efficacy evaluation were used to calculate a total score. 22 questions are divided among 4 subscales: Rhinologic (7 questions), Ear/Facial Symptoms (4 questions), Sleep Function (3 questions), and Psychological Issues (6 questions). Each item was rated on the 5-point scale. The total score can range from 0-110, 0 being the best and 110 being the worst.
  0: No problem
  1. Very mild problem
  2. Mild or slight problem
  3. Moderate problem
  4. Severe problem
  5. Problem as bad as can be Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  units on a scale
    number analyzed (Participants) | 82 | 80 | 80 | 77 | 319
    (all) | 53.7 [14 to 95] | 46.1 [14 to 95] | 51.8 [0 to 108] | 52.4 [6 to 103] | 51 [0 to 108]
Medical Outcomes Study Sleep Scale Revised (MOS Sleep-R) [Mean (Full Range); unit: units on a scale] — The MOS Sleep-R is a brief, self-administered, validated questionnaire designed to measure key aspects of sleep, such as disturbance, adequacy, somnolence, and quantity. The 12-item version with a 4-week recall was used in this study. The score range for the 12-item version is 0 to 100, lower scores indicating better sleep and higher scores indicating worse sleep. The scale yields a Sleep Problem Index and scores on the following 6 subscales: Sleep Disturbance, Snoring, Shortness of Breath or Headache, Sleep Adequacy, Sleep Somnolence, and Sleep Quantity. Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  units on a scale
    number analyzed (Participants) | 82 | 81 | 80 | 79 | 322
    (all) | 42.8 [5.6 to 97.2] | 37.8 [2.8 to 77.8] | 46.6 [11.1 to 91.7] | 43.7 [11.1 to 88.9] | 42.71 [2.8 to 97.2]
Rhinosinusitis Disability Index (RSDI) Total Score [Mean (Full Range); unit: units on a scale] — The RSDI is a subject-completed instrument that evaluates the self-perceived impact of disease specific head and neck disorders. The RSDI has 30 items in 3 domains: Physical (11 items), Functional (9 items), and Emotional (10 items). The RSDI scale ranges from 0-120, 0 being better quality of life and less impact of CRS on daily function and 120 being worse quality of life and more impact of CRS on daily function. Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  units on a scale
    number analyzed (Participants) | 82 | 80 | 79 | 78 | 319
    (all) | 48.3 [2 to 120] | 39.8 [2 to 96] | 45.2 [3 to 91] | 45.4 [5 to 117] | 44.69 [2 to 120]
Short Form (36) Health Survey Version 2 (SF-36v2) - Mental Component [Mean (Full Range); unit: units on a scale] — The SF-36v2 is a multipurpose, scaled, 36-item, subject-completed validated questionnaire that measures 8 domains of health: limitations in physical activities, limitations in social activities, limitations in usual role activities, bodily pain, general mental health, limitations in usual role activities, vitality, and general health. It yields scale scores for each of the 8 health domains, and 2 summary measures of physical and mental health. Each scale range is from 0-100. A lower score means more disability and a higher score means less disability. Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  units on a scale
    number analyzed (Participants) | 82 | 81 | 79 | 79 | 321
    (all) | 47.6 [23.66 to 63.99] | 49.0 [22.18 to 63.08] | 46.0 [18.06 to 58.7] | 47.8 [15.26 to 62.61] | 47.6 [15.26 to 63.99]
Short Form (36) Health Survey Version 2 (SF-36v2) - Physical Component [Mean (Full Range); unit: units on a scale] — The SF-36v2 is a multipurpose, scaled, 36-item, subject-completed validated questionnaire that measures 8 domains of health: limitations in physical activities, limitations in social activities, limitations in usual role activities, bodily pain, general mental health, limitations in usual role activities, vitality, and general health perceptions. It yields scale scores for each of the 8 health domains, and 2 summary measures of physical and mental health. Each scale range is from 0-100. A lower score means more disability and a higher score means less disability. Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  units on a scale
    number analyzed (Participants) | 82 | 81 | 79 | 79 | 321
    (all) | 43.5 [27.75 to 57.53] | 44.7 [28.01 to 60.58] | 43.9 [28.36 to 60.91] | 43.9 [22.58 to 59.26] | 44 [22.58 to 60.91]
Peak Nasal Inspiratory Flow (PNIF) [Mean (Full Range); unit: L/min] — The PNIF is an assessment of nasal passage obstruction and was measured using an In-Check portable nasal inspiratory flow meter. To measure PNIF, a mask was placed over the nose during inspiration and inspiratory flow was recorded. Each subject inhaled 3 times and each measurement was recorded. The PNIF value used was the greatest of the 3 results at each time point. Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  L/min
    number analyzed (Participants) | 82 | 81 | 79 | 79 | 321
    (all) | 105.1 [30 to 350] | 111.6 [0 to 360] | 97.1 [30 to 350] | 103.2 [25 to 340] | 104.3 [0 to 360]
Nasal Polyp Surgery Eligibility [Count of Participants; unit: Participants] — Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  Participants
    number analyzed (Participants) | 82 | 81 | 80 | 78 | 321
    (all) | 53 | 45 | 44 | 47 | 189

OUTCOME MEASURES:

1. Primary Outcome: Change in 7-day Average Instantaneous Morning Diary Congestion/Obstruction Symptoms
Description: Subjects reported nasal symptoms using the electronic diary twice daily immediately before dosing.
  0: None
  1. Mild, symptoms clearly present, but minimal awareness, and easily tolerated
  2. Moderate, definite awareness of symptoms that is bothersome but tolerable
  3. Severe, symptoms that are hard to tolerate, cause interference with activities or daily living
  The change from baseline in instantaneous morning diary symptom scores averaged over 7 days prior to the Week 4 Visit of the double-blind treatment phase
Time Frame: Baseline, Week 4 of the double-blind treatment phase
Population: Missing data were imputed using the multiple imputation method in the primary analyses for the co-primary efficacy variables. For other efficacy analyses, missing or invalid values were not imputed.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Matching Placebo Twice Daily x 16 weeks, then OPN-375 400 μg (open-label) BID x 8 weeks
Arm/Group | Placebo | OPN-375 100 μg BID | OPN-375 200 μg BID | OPN-375 400 μg BID
Number analyzed (Participants) | 77 | 78 | 79 | 78
units on a scale | -0.26 (0.08) | -0.53 (0.08) | -0.56 (0.08) | -0.67 (0.08)

2. Primary Outcome: Change in Total Polyp Grade
Description: Polyp grading of each nasal cavity was determined by a nasal polyp grading scale score measured by nasoendoscopy. A summary of the changes from baseline to Week 16 in total polyp grade.
  0: No polyps
  1. Mild polyposis: polyps not reaching below the inferior border of the middle turbinate
  2. Moderate polyposis: polyps reaching below the inferior border of the middle concha, but not the inferior border of the inferior turbinate
  3. Severe polyposis large polyps reaching below the lower inferior border of the inferior turbinate
  Reduction in total polyp grade (sum of scores from both nasal cavities) at Week 16 of double-blind treatment phase; Included patients with nasal polyps at baseline
Time Frame: Baseline, Week 16 of the double-blind treatment phase
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | OPN-375 100 μg BID | OPN-375 200 μg BID | OPN-375 400 μg BID
Number analyzed (Participants) | 68 | 75 | 68 | 75
units on a scale | -0.57 (0.14) | -1.04 (0.14) | -1.14 (0.14) | -1.14 (0.14)

3. Secondary Outcome: Congestion/Obstruction Scores (7-day Instantaneous Morning)
Description: Subjects reported nasal symptoms using the electronic diary twice daily immediately before dosing.
  0: None
  1. Mild, symptoms clearly present, but minimal awareness, and easily tolerated
  2. Moderate, definite awareness of symptoms that is bothersome but tolerable
  3. Severe, symptoms that are hard to tolerate, cause interference with activities or daily living
  The change from baseline in instantaneous morning diary symptom scores averaged over 7 days prior to the Week 16 Visit of the double-blind treatment phase
Time Frame: Baseline, Week 16 of the double-blind treatment phase
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Groups:
- OPN-375 100 μg Twice Daily: 100 μg Twice Daily x 16 weeks, then OPN-375 400 μg (open-label) BID x 8 weeks
- OPN-375 200 μg Twice Daily: 200 μg Twice Daily x 16 weeks, then OPN-375 400 μg (open-label) BID x 8 weeks
- OPN-375 400 μg Twice Daily: OPN-375 400 μg Twice Daily x 16 weeks, then OPN-375 400 μg (open-label) BID x 8 weeks
Arm/Group | Placebo | OPN-375 100 μg Twice Daily | OPN-375 200 μg Twice Daily | OPN-375 400 μg Twice Daily
Number analyzed (Participants) | 82 | 81 | 80 | 79
units on a scale | -0.53 (0.11) | -0.93 (0.10) | -0.99 (0.10) | -1.07 (0.10)

4. Secondary Outcome: Change in Rhinorrhea Score (7-day Instantaneous Morning)
Description: as for outcome 3
Time Frame: Baseline, Week 16 of the double-blind treatment phase
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | OPN-375 100 μg BID | OPN-375 200 μg BID | OPN-375 400 μg BID
Number analyzed (Participants) | 82 | 81 | 80 | 79
units on a scale | -0.50 (0.10) | -0.80 (0.10) | -0.89 (0.10) | -0.92 (0.10)

5. Secondary Outcome: Facial Pain or Pressure Score (7-day Instantaneous Morning)
Description: as for outcome 3
Time Frame: Baseline, Week 16 of the double-blind treatment phase
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | OPN-375 100 μg BID | OPN-375 200 μg BID | OPN-375 400 μg BID
Number analyzed (Participants) | 82 | 81 | 80 | 79
units on a scale | -0.41 (0.11) | -0.65 (0.10) | -0.72 (0.10) | -0.68 (0.10)

6. Secondary Outcome: Hyposmia Score (7-day Instantaneous Morning)
Description: as for outcome 3
Time Frame: Baseline, Week 16 of the double-blind treatment phase
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | OPN-375 100 μg BID | OPN-375 200 μg BID | OPN-375 400 μg BID
Number analyzed (Participants) | 82 | 81 | 80 | 79
units on a scale | -0.23 (0.12) | -0.45 (0.11) | -0.53 (0.11) | -0.60 (0.11)

7. Secondary Outcome: Sinonasal Outcome Test 22 (SNOT-22) Total Score
Description: SNOT-22 is a subject-completed questionnaire that consists of 22 questions. The questions on the SNOT-22 efficacy evaluation were used to calculate a total score. 22 questions are divided among 4 subscales: Rhinologic (7 questions), Ear/Facial Symptoms (4 questions), Sleep Function (3 questions), and Psychological Issues (6 questions). Each item was rated on the 5-point scale. The total score can range from 0-110, 0 being the best and 110 being the worst.
  0: No problem
  1. Very mild problem
  2. Mild or slight problem
  3. Moderate problem
  4. Severe problem
  5. Problem as bad as it can be
Time Frame: Baseline, Week 16 of the double-blind treatment phase, Week 24 of the end of open-label treatment phase
Population: Number of patients analyzed at Week 24 is lower as some patients elected not to participate in the open-label extension phase or withdrew during the open-label extension phase.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | OPN-375 100 μg BID | OPN-375 200 μg BID | OPN-375 400 μg BID
Number analyzed (Participants) | 82 | 80 | 80 | 77
units on a scale
  Change from baseline to Week 16 | -10.96 (2.07) | -18.32 (2.05) | -19.56 (2.04) | -19.80 (2.05)
  Change from baseline to Week 24 (all pts on 400 μg: number analyzed (Participants) | 62 | 69 | 64 | 69
  Change from baseline to Week 24 (all pts on 400 μg | -20.78 (2.10) | -21.20 (2.07) | -23.28 (2.08) | -21.72 (2.07)

8. Secondary Outcome: MOS Sleep-R Score
Description: The MOS Sleep-R is a brief, self-administered, validated questionnaire designed to measure key aspects of sleep, such as disturbance, adequacy, somnolence, and quantity. The 12-item version with a 4-week recall was used in this study. The score range for the 12-item version is 0 to 100, lower scores indicating better sleep and higher scores indicating worse sleep. The scale yields a Sleep Problem Index and scores on the following 6 subscales: Sleep Disturbance, Snoring, Shortness of Breath or Headache, Sleep Adequacy, Sleep Somnolence, and Sleep Quantity.
Time Frame: Baseline, Week 16 of the double-blind treatment phase
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | OPN-375 100 μg BID | OPN-375 200 μg BID | OPN-375 400 μg BID
Number analyzed (Participants) | 82 | 81 | 80 | 79
units on a scale | -8.53 (1.61) | -10.96 (1.59) | -14.24 (1.59) | -10.66 (1.55)

9. Secondary Outcome: Rhinosinusitis Disability Index (RSDI) Total Score
Description: The RSDI is a subject-completed instrument that evaluates the self-perceived impact of disease specific head and neck disorders. The RSDI has 30 items in 3 domains: Physical (11 items), Functional (9 items), and Emotional (10 items). The RSDI scale ranges from 0-120, 0 being better quality of life and less impact of CRS on daily function and 120 being worse quality of life and more impact of CRS on daily function.
Time Frame: Baseline, Week 16 of the double-blind treatment phase
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | OPN-375 100 μg BID | OPN-375 200 μg BID | OPN-375 400 μg BID
Number analyzed (Participants) | 67 | 71 | 69 | 73
units on a scale | -10.71 (2.07) | -17.08 (1.99) | -16.44 (2.02) | -16.37 (1.94)

10. Secondary Outcome: SF-36v2 - Mental Component
Description: The SF-36v2 is a multipurpose, scaled, 36-item, subject-completed validated questionnaire that measures 8 domains of health: limitations in physical activities, limitations in social activities, limitations in usual role activities, bodily pain, general mental health, limitations in usual role activities, vitality, and general health. It yields scale scores for each of the 8 health domains, and 2 summary measures of physical and mental health. Each scale range is from 0-100. A lower score means more disability and a higher score means less disability.
Time Frame: Baseline, Week 16 of the double-blind treatment phase, Week 24 of the end of open-label treatment phase
Population: as for outcome 7
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | OPN-375 100 μg BID | OPN-375 200 μg BID | OPN-375 400 μg BID
Number analyzed (Participants) | 68 | 74 | 70 | 75
units on a scale
  Week 16 | 0.70 (0.87) | 3.19 (0.84) | 4.03 (0.85) | 1.83 (0.82)
  Week 24 (all pts on 400 μg OPN-375 BID wks 17-24): number analyzed (Participants) | 64 | 69 | 63 | 71
  Week 24 (all pts on 400 μg OPN-375 BID wks 17-24) | 4.44 (0.83) | 3.37 (0.80) | 5.82 (0.84) | 3.61 (0.78)

11. Secondary Outcome: SF-36v2 - Physical Component
Description: The SF-36v2 is a multipurpose, scaled, 36-item, subject-completed validated questionnaire that measures 8 domains of health: limitations in physical activities, limitations in social activities, limitations in usual role activities, bodily pain, general mental health, limitations in usual role activities, vitality, and general health perceptions. It yields scale scores for each of the 8 health domains, and 2 summary measures of physical and mental health. Each scale range is from 0-100. A lower score means more disability and a higher score means less disability.
Time Frame: Baseline, Week 16 of the double-blind treatment phase, Week 24 of the end of open-label treatment phase
Population: as for outcome 7
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | OPN-375 100 μg BID | OPN-375 200 μg BID | OPN-375 400 μg BID
Number analyzed (Participants) | 68 | 74 | 70 | 75
units on a scale
  Week 16 | 2.67 (0.76) | 4.12 (0.74) | 5.19 (0.74) | 3.58 (0.72)
  Week 24 (all pts on 400 μg OPN-375 BID wks 17-24): number analyzed (Participants) | 64 | 69 | 63 | 71
  Week 24 (all pts on 400 μg OPN-375 BID wks 17-24) | 6.97 (0.78) | 6.55 (0.75) | 7.18 (0.78) | 4.90 (0.73)

12. Secondary Outcome: Patient Global Impression of Change (PGIC) Score
Description: Subject responses to the question: "Since starting the study drug, how would you rate the change in your symptoms?" Percentage includes patients who scored either "very much improved," "much improved," or "minimally improved."
Time Frame: Week 16 of the double-blind treatment phase, Week 24 of the end of open-label treatment phase
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | OPN-375 100 μg BID | OPN-375 200 μg BID | OPN-375 400 μg BID
Number analyzed (Participants) | 68 | 73 | 70 | 75
Participants
  Week 16 | 51 | 56 | 62 | 67
  Week 24 (all pts on 400 μg OPN-375 BID wks 17-24) | 59 | 62 | 62 | 66

13. Secondary Outcome: Peak Nasal Inspiratory Flow (PNIF)
Description: The PNIF is an assessment of nasal passage obstruction and was measured using an In-Check portable nasal inspiratory flow meter. To measure PNIF, a mask was placed over the nose during inspiration and inspiratory flow was recorded. Each subject inhaled 3 times and each measurement was recorded. The PNIF value used was the greatest of the 3 results at each time point.
Time Frame: Baseline, Week 16 of the double-blind treatment phase, Week 24 of the open-label treatment phase
Population: as for outcome 7
Measure: Least Squares Mean (Standard Deviation); unit: L/min
Arm/Group | Placebo | OPN-375 100 μg BID | OPN-375 200 μg BID | OPN-375 400 μg BID
Number analyzed (Participants) | 68 | 75 | 70 | 74
L/min
  Week 16 | 17.26 (6.15) | 36.57 (6.06) | 35.94 (6.08) | 35.43 (5.95)
  Week 24 (all pts on 400 μg OPN-375 BID wks 17-24): number analyzed (Participants) | 64 | 70 | 63 | 71
  Week 24 (all pts on 400 μg OPN-375 BID wks 17-24) | 34.92 (6.31) | 41.61 (6.21) | 44.70 (6.27) | 35.64 (6.09)

14. Secondary Outcome: Polyp Grade of 0 in at Least One Nostril
Description: Polyp grading of each nasal cavity was determined by a nasal polyp grading scale score measured by nasoendoscopy. This outcome measured how many patients with a polyp grad of 0 in at least 1 nostril.
  0: No polyps
  1. Mild polyposis: polyps not reaching below the inferior border of the middle turbinate
  2. Moderate polyposis: polyps reaching below the inferior border of the middle concha, but not the inferior border of the inferior turbinate
  3. Severe polyposis large polyps reaching below the lower inferior border of the inferior turbinate
Time Frame: Baseline, Week 16 of the double-blind treatment phase, Week 24 of the end of open-label treatment phase
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Groups:
- OPN-375 400 μg Twice Daily: 400 μg Twice Daily x 16 weeks, then OPN-375 400 μg (open-label) BID x 8 weeks
Arm/Group | Placebo | OPN-375 100 μg Twice Daily | OPN-375 200 μg Twice Daily | OPN-375 400 μg Twice Daily
Number analyzed (Participants) | 68 | 75 | 68 | 75
Participants
  Week 16 | 9 | 19 | 12 | 14
  Week 24 (all pts on 400 μg OPN-375 BID wks 17-24): number analyzed (Participants) | 64 | 70 | 64 | 71
  Week 24 (all pts on 400 μg OPN-375 BID wks 17-24) | 17 | 24 | 16 | 19

15. Secondary Outcome: Nasal Polyp Surgery Eligilbilty
Description: A subject was considered eligible for surgical intervention if the following conditions were met:
  * Subject has had moderate symptoms of congestion from nasal polyposis for ≥ 3 months.
  * Subject continues to suffer from at least moderate symptoms despite use of topical steroids at conventional doses for ≥ 6 weeks.
  * Subject continues to suffer from at least moderate symptoms despite use (or previous use) of saline lavage for ≥ 6 weeks.
  * Subject has endoscopically visualized bilateral nasal polyposis of at least moderate severity (nasal polyp grading score ≥ 2 in at least 1 nostril).
Time Frame: Baseline, Week 16 of the double-blind treatment phase, Week 24 of the open-label extension phase
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 100 μg OPN-375 | 200 μg OPN-375 | 400 μg EDS-FLU
Number analyzed (Participants) | 68 | 74 | 69 | 75
Participants
  Week 16 | 27 | 17 | 21 | 19
  Week 24 (all pts on OPN-375 400 mcg BID wks 17-24): number analyzed (Participants) | 64 | 70 | 63 | 70
  Week 24 (all pts on OPN-375 400 mcg BID wks 17-24) | 15 | 14 | 17 | 16

ADVERSE EVENTS:
Description: The Safety Analysis Set (SAS) included all ITT subjects who received at least 1 dose of study drug. The SAS was used for the analysis of safety. The treatment group classification in the SAS was according to the treatment actually received.
Groups:
- Placebo (Double-Blind Phase): 100 μg BID or 200 μg BID or 400 μg Matching Placebo BID x 16 weeks
- OPN-375 100 μg BID (Double-Blind Phase): OPN-375 100 μg BID x 16 weeks
- OPN-375 200 μg BID (Double-Blind Phase): OPN-375 200 μg BID x 16 weeks
- OPN-375 400 μg BID (Double-Blind Phase): OPN-375 400 μg BID x 16 weeks
- OPN-375 400 μg (Open-Label Phase): OPN-375 400 μg BID x 8 weeks
Arm/Group | Placebo (Double-Blind Phase) | OPN-375 100 μg BID (Double-Blind Phase) | OPN-375 200 μg BID (Double-Blind Phase) | OPN-375 400 μg BID (Double-Blind Phase) | OPN-375 400 μg (Open-Label Phase)
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/81 | 0/80 | 0/79 | 0/282
Serious Adverse Events (participants affected / at risk) | 0/82 | 1/81 | 0/80 | 1/79 | 2/282
Other Adverse Events (participants affected / at risk) | 42/82 | 40/81 | 45/80 | 50/79 | 38/282
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Double-Blind Phase) (N=82) | OPN-375 100 μg BID (Double-Blind Phase) (N=81) | OPN-375 200 μg BID (Double-Blind Phase) (N=80) | OPN-375 400 μg BID (Double-Blind Phase) (N=79) | OPN-375 400 μg (Open-Label Phase) (N=282)
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Double-Blind Phase) (N=82) | OPN-375 100 μg BID (Double-Blind Phase) (N=81) | OPN-375 200 μg BID (Double-Blind Phase) (N=80) | OPN-375 400 μg BID (Double-Blind Phase) (N=79) | OPN-375 400 μg (Open-Label Phase) (N=282)
Ear Pain (Ear and labyrinth disorders) | 1 | 2 | 0 | 0 | 1
Cataract Nuclear (Eye disorders) | 2 | 1 | 0 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Acute Sinusitis (Infections and infestations) | 4 | 5 | 6 | 8 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 7 | 1 | 4 | 5 | 2
Nasopharyngitis (Infections and infestations) | 4 | 3 | 2 | 4 | 3
Bronchitis (Infections and infestations) | 2 | 2 | 2 | 3 | 0
Influenza (Infections and infestations) | 3 | 2 | 2 | 2 | 0
Pharyngitis (Infections and infestations) | 2 | 0 | 1 | 3 | 0
Otitis Media (Infections and infestations) | 1 | 2 | 0 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Weight Increased (Investigations) | 0 | 0 | 2 | 0 | 0
Intraocular Pressure Increased (Investigations) | 2 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 2 | 2 | 0 | 2
Epistaxis (Spontaneously Reported by Subject) (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 7 | 6 | 12
Nasal Mucosal Disorder (Respiratory, thoracic and mediastinal disorders) | 5 | 11 | 6 | 6 | 1
Nasal Septal Ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 5 | 4 | 5
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2 | 6 | 1
Nasal Septum Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 3 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1 | 3 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0
Epistaxis (Found on Nasoendoscopy) (Respiratory, thoracic and mediastinal disorders) | 3 | 8 | 9 | 13 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure agreement is described in CTA between sponsor and PI